CLINICAL TRIAL: NCT06908265
Title: Clinical Evaluation of the Antibacterial Activity of Thioglycosides Extracted from White Mustard - Bamberka in Oral Hygiene.
Brief Title: Clinical Evaluation of the Antibacterial Activity of Thioglycosides Extracted from White Mustard - Bamberka in Oral Hygiene. Evaluation of Periodontal Parameters and Oral Microbiota in Patients.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KB/58/2011
Record Dates: First submitted 2025-03-19; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Gingival and Periodontal Disease; Caries, Dental
Keywords: Caries.; thioglycosides; periodontitis; gingivitis; lactobacillus; toothpaste; mustard
MeSH Terms: conditions — Periodontal Diseases; Dental Caries; Periodontitis; Gingivitis

STUDY DESIGN:
Intervention Model Description: Participants were divided into two groups, experimental and control. The experimental group received an intervention - mustard toothpaste. The control group received a control toothpaste without mustard extract.
Who Masked: Participant, Investigator
Masking Description: Participants were randomly assigned to two groups and blinded - Experimental vs placebo. They got toothpaste samples in identically marked white tubes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Participants in this group receive a herbal toothpaste containing white mustard (Sinapis alba) extract.
  The toothpaste is formulated with 0.5% white mustard extract, known for its antibacterial properties.
  Participants are instructed to brush their teeth twice daily for 4 weeks using this toothpaste.
  The primary goal is to evaluate its effect on plaque index (PI), approximal plaque index (API), gingival index (GI), bleeding on probing (BoP), and the bacterial loads of Streptococcus mutans and Lactobacillus spp.
  Interventions: Drug: Toothpaste including mustard extract
- Control Group (Placebo Comparator): Participants in this group receive a placebo toothpaste, which has the same base formulation as the experimental toothpaste but without white mustard extract.
  They are also instructed to brush their teeth twice daily for 4 weeks using the assigned toothpaste.
  This arm serves as a control group to compare the effects of the herbal toothpaste with a non-herbal alternative.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Toothpaste including mustard extract — Intervention: Herbal toothpaste containing 0.5% white mustard (Sinapis alba) extract. To assess its effect on plaque index (PI), approximal plaque index (API), gingival index (GI), bleeding on probing (BoP), and bacterial loads of Streptococcus mutans and Lactobacillus spp.
  Dosage and Usage: Participants brush their teeth twice daily for 4 weeks with the assigned toothpaste.
  Arms: Experimental Group
Drug: Placebo — lacebo toothpaste, formulated identically to the experimental toothpaste but without white mustard extract. Serves as a control to compare the antibacterial and clinical effects of the herbal toothpaste.
  Dosage and Usage: Participants brush their teeth twice daily for 4 weeks with the placebo toothpaste.
  Arms: Control Group

SUMMARY:
Brief Summary

The goal of this randomized clinical trial is to evaluate the clinical and antibacterial effects of a herbal toothpaste containing white mustard (Sinapis alba) extract in patients diagnosed with gingivitis. The main questions it aims to answer are:

Does the herbal toothpaste significantly reduce plaque index (PI), approximal plaque index (API), gingival index (GI), and bleeding on probing (BoP) compared to a placebo toothpaste?

Does the herbal toothpaste effectively reduce the bacterial loads of Streptococcus mutans and Lactobacillus spp. in saliva compared to a placebo?

Researchers will compare the effects of the herbal toothpaste to a placebo toothpaste to determine its efficacy in improving periodontal parameters and reducing bacterial levels.

Participants will:

Be randomly assigned to one of two groups: test group (herbal toothpaste) or control group (placebo toothpaste).

Use the assigned toothpaste twice daily for 4 weeks.

Undergo clinical evaluations at baseline (T0) and after 4 weeks (T1), including measurements of PI, API, GI, and BoP.

Provide saliva samples at T0 and T1 for microbiological analysis of Streptococcus mutans and Lactobacillus spp. bacterial loads.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years,
* the presence of at least 20 teeth excluding third molars,
* a diagnosis of gingivitis according to the 2017 World Workshop
* non-smokers.
* the motivation to take part in the study,
* proper oral home hygiene
* sign a consent agreement for the participation in the study

Exclusion Criteria:

* patients aged <18
* the presence of less than 20 teeth
* severe systemic diseases and diseases that require regular systemic drugs (diabetes mellitus)
* the use of systemic antibiotics during the last 3 months or local antiseptics that may affect biofilm formation (antibacterial mouth rinses containing chlorhexidine 4 weeks or less prior recruitment)
* allergy to mustard or any other compound of experimental toothpaste
* patients undergoing orthodontic treatment
* women who were pregnant or breastfeeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change in Plaque Index (PI) from Baseline (T0) to Week 4 (T1) | From start of intervention, 4 weeks to end of intervention and data collection.
  Change in Plaque Index (PI) from Baseline (T0) to Week 4 (T1) Measured using the Silness and Loe Plaque Index (PI) Scale to assess plaque accumulation on tooth surfaces.
  Unit: Plaque score (0-3 scale). Time Frame: Baseline (T0) and Week 4 (T1).
Change in Bleeding on Probing (BoP) from Baseline (T0) to Week 4 (T1) | From start of intervention, 4 weeks to end of intervention and data collection.
  Change in Bleeding on Probing (BoP) from Baseline (T0) to Week 4 (T1) Measured using the Ainamo and Bay method, which evaluates gingival bleeding after gentle probing. Unit: Percentage of bleeding sites. Time Frame: Baseline (T0) and Week 4 (T1).

SECONDARY OUTCOMES:
Change in Approximal Plaque Index (API) from Baseline (T0) to Week 4 (T1) | 4 weeks
  Measured based on the presence of plaque in interdental areas. Unit: Percentage of interdental sites with plaque. Time Frame: Baseline (T0) and Week 4 (T1).
Change in Gingival Index (GI) from Baseline (T0) to Week 4 (T1) | 4 weeks
  Measured using the Loe and Silness Gingival Index (GI) Scale to assess the degree of gingival inflammation.
  Unit: Gingival index score (0-3 scale). Time Frame: Baseline (T0) and Week 4 (T1).
Change in Salivary Bacterial Loads of Streptococcus mutans and Lactobacillus spp. from Baseline (T0) to Week 4 (T1) | 4 weeks
  Measured using the Caries Risk Test (CRT, Ivoclar Vivadent) to determine bacterial colony counts in saliva samples.
  Unit: Colony-forming units per milliliter (CFU/ml). Time Frame: Baseline (T0) and Week 4 (T1).

IPD SHARING:
Plan to Share IPD: Yes
We will share data including results and statistical analyses in publication after the complement od the study.
Supporting Information: Study Protocol
Time Frame: The publication will be available in open-access journal

REFERENCES:
- [Background] Arweiler NB, Pergola G, Kuenz J, Hellwig E, Sculean A, Auschill TM. Clinical and antibacterial effect of an anti-inflammatory toothpaste formulation with Scutellaria baicalensis extract on experimental gingivitis. Clin Oral Investig. 2011 Dec;15(6):909-13. doi: 10.1007/s00784-010-0471-1. Epub 2010 Oct 9. PMID 20936314
- [Background] Melrose J. The Glucosinolates: A Sulphur Glucoside Family of Mustard Anti-Tumour and Antimicrobial Phytochemicals of Potential Therapeutic Application. Biomedicines. 2019 Aug 19;7(3):62. doi: 10.3390/biomedicines7030062. PMID 31430999
- [Background] David JR, Ekanayake A, Singh I, Farina B, Meyer M. Effect of white mustard essential oil on inoculated Salmonella sp. in a sauce with particulates. J Food Prot. 2013 Apr;76(4):580-7. doi: 10.4315/0362-028X.JFP-12-375. PMID 23575118
- [Background] Eichel V, Schuller A, Biehler K, Al-Ahmad A, Frank U. Antimicrobial effects of mustard oil-containing plants against oral pathogens: an in vitro study. BMC Complement Med Ther. 2020 May 24;20(1):156. doi: 10.1186/s12906-020-02953-0. PMID 32448381